CLINICAL TRIAL: NCT05785923
Title: The Impact of Point-of-Care Ultrasound Echocardiography on the Disposition of Low-Risk Chest Pain Patients in the Emergency Department
Brief Title: Low-Risk Chest Pain Echo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Adrienne Malik, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00149603
Record Dates: First submitted 2023-02-13; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echo Arm (Experimental): Chest pain patients identified by their treating physician as being low-risk chest pain will undergo a point-of-care echocardiogram performed by a trained emergency medicine attending or resident prior to discharge from the emergency department. The physician of record will review this ultrasound and it will be documented whether the findings on the ultrasound changed the physician of record's disposition decision for the patient or the follow up instructions or medications.
  Interventions: Diagnostic Test: Point-of-Care Echocardiogram
- Usual Care (No Intervention): Chest pain patients identified by their treating physician as being low-risk chest pain will receive the usual care for their condition.

INTERVENTIONS:
Diagnostic Test: Point-of-Care Echocardiogram — Four view ultrasound of the heart performed at the bedside by trained emergency medicine physicians.
  Arms: Echo Arm

SUMMARY:
Pilot study to assess if a bedside point-of-care echocardiogram performed on emergency department patients identified as low-risk chest pain prior to discharge significantly changes patient disposition or follow up instructions.

ELIGIBILITY:
Inclusion Criteria:

* Adults presenting to the emergency department with an isolated chief complaint of chest pain with a HEART score of 3 or less
* Emergency physician of record has decided to discharge this patient from the Emergency Department

Exclusion Criteria:

* Patients who are unable to consent for themselves
* History of cardiac transplant or LVAD
* Pediatric patients
* Patients presenting with multiple complaints in addition to chest pain
* Echocardiogram already performed on patient during usual care
* Patients with another non-cardiac admittable diagnosis
* HEART score greater than or equal to 4

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-05 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Disposition | Day of enrollment
  Will assess if the result of the point-of-care echocardiogram resulted in the physician of record changing subject disposition from discharge to admission. We will assess this by asking the physician of record what the disposition plan is for the patient and recording their answer on IRB approved data collection sheet.

SECONDARY OUTCOMES:
Follow up instructions | day of enrollment
  Will assess if the result of the point-of-care echocardiogram changed the follow up instructions or discharge medication decision for the enrolled subject as determined by the physician of record by asking them if the echo results caused them to add any additional discharge instructions for the patient. We will record their answer on the IRB approved data collection sheet.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laureano-Phillips J, Robinson RD, Aryal S, Blair S, Wilson D, Boyd K, Schrader CD, Zenarosa NR, Wang H. HEART Score Risk Stratification of Low-Risk Chest Pain Patients in the Emergency Department: A Systematic Review and Meta-Analysis. Ann Emerg Med. 2019 Aug;74(2):187-203. doi: 10.1016/j.annemergmed.2018.12.010. Epub 2019 Feb 2. PMID 30718010
- [Background] Rainer TH, Leung YK, Lee A, Chan PY, Cheng NM, Wong JK, Yan BP, Ahuja AT, Graham CA. Add-on tests for improving risk-stratification in emergency department patients with chest pain who are at low to moderate risk of 30-day major adverse cardiac events. Int J Cardiol. 2016 Oct 1;220:299-306. doi: 10.1016/j.ijcard.2016.05.057. Epub 2016 May 14. PMID 27390945
- [Background] Guner NG, Yurumez Y, Yucel M, Alacam M, Guner ST, Ercan B. Effects of Point-of-care Ultrasonography on the Diagnostic Process of Patients Admitted to the Emergency Department with Chest Pain: A Randomised Controlled Trial. J Coll Physicians Surg Pak. 2020 Dec;30(12):1262-1268. doi: 10.29271/jcpsp.2020.12.1262. PMID 33397050
- [Background] Buhumaid RE, St-Cyr Bourque J, Shokoohi H, Ma IWY, Longacre M, Liteplo AS. Integrating point-of-care ultrasound in the ED evaluation of patients presenting with chest pain and shortness of breath. Am J Emerg Med. 2019 Feb;37(2):298-303. doi: 10.1016/j.ajem.2018.10.059. Epub 2018 Oct 30. PMID 30413369